CLINICAL TRIAL: NCT06708689
Title: Retrospective Case-control Study of Central Line Botriomycoma in Children on Home Parenteral Nutrition: Epidemiology, Risk Factors, Treatments
Brief Title: Overview of Botriomycoma in Children with a Central Line: Epidemiology, Risk Factors, Treatments
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0638
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Home Parenteral Nutrition; Intestinal Failure; Central Line; Botriomycoma; Infection; Sepsis; Antibiotics
MeSH Terms: conditions — Intestinal Failure; Infections; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Case / patients: Pediatric patients requiring a long-term central line for home parenteral nutrition:
  * home parenteral nutrition patients
  * diagnosed with at least on episode of botriomycoma on their central line
  * 0 to 18 years of age at diagnosis of botriomycoma
- Control: Pediatric patients requiring a long-term central line for home parenteral nutrition:
  * home parenteral nutrition patients
  * never diagnosed with an episode of botriomycoma on their central line
  * 0 to 18 years of age at diagnosis

SUMMARY:
Botriomycomas are frequent benign tumors in children. Their appearance on the central catheter orifice is a known event in clinical practice, but one that has been little studied. This lesion could lead to changes in pathways and an increase in the number of sepsis events, which would promote thrombosis and thus depletion of venous capital in patients who have been dependent on a central line for many years.

This study is a pilot study which will enable us to better identify the risk factors for the development of such a tumour, and to take stock of the different treatments used and their respective efficacy.

ELIGIBILITY:
Inclusion Criteria:

* home parenteral nutrition patients
* never diagnosed with an episode of botriomycoma on their central line
* 0 to 18 years of age at diagnosis

Exclusion Criteria:

* Botriomycoma more than 10 years old at time of data collection (or lack of data)
* Patient over 18 years of age
* Not on home parenteral nutrition patients

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with intestinal failures requiring a long-term central line for home parenteral nutrition in France
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Appearance of Botryomycoma | From first diagnosis through a follow-up period of 2 years.
  genetic characteristics (origin, phototype), local factors (mechanical, infectious), and general factors (history of sepsis).
Recurrence of Botryomycoma | From first diagnosis through a follow-up period of 2 years.
  analyze risk factors for recurrence and evolution under different treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Mère-Enfant, Bron, France